CLINICAL TRIAL: NCT04719871
Title: Rate of Visual Field Progression Before and After Posterior Vitreous Detachment
Brief Title: Vitreous Detachment and Glaucoma Progression
Acronym: REVEAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0696
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Glaucoma; Posterior Vitreous Detachment
Keywords: Glaucoma; Vitreous; Progression
MeSH Terms: conditions — Glaucoma; Vitreous Detachment; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with posterior vitreous detachment: patient with stage 3 or more of posterior vitreous detachment on optical coherence tomography
- without posterior vitreous detachment: patient with stage 2 or less of posterior vitreous detachment on optical coherence tomography

SUMMARY:
Posterior vitreous detachment is a common event. With optical coherence tomography, the investigators can precisely follow the stage of posterior vitrous detachment. In this study, the investigators investigate if the loss of contact between the vitreous and the fovea is the start of glaucoma progression.

ELIGIBILITY:
Inclusion criteria:

* Patient with glaucoma
* at least 4 years of follow up
* at least 6 visual fields
* at least 4 optical coherence tomographies

Exclusion criteria:

* pars plana vitrectomy
* others ophtalmological or neurological disease which can modify visual fields

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective cohort of patient with glaucoma follow in Montpellier hospital
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Glaucoma progression | 1 day
  glaucoma progression based on analysis of visual fields

SECONDARY OUTCOMES:
RNFL decr | 1 day
  slope of decrease

CONTACTS AND LOCATIONS:
Overall Officials: MAX VILLAIN, PHD, Study Director — UH MONTPELLIER
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC